CLINICAL TRIAL: NCT01707524
Title: Effect of Left Versus Right Radial Artery Access on Radiation Exposure in Patients With Predictors of Potential Trans-radial Access Failure
Brief Title: Left Versus Right Radial Artery and Radiation Exposure in Patients With Predictors of Trans-radial Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Principal Investigator, John Coppola, Assistant Professor of Medicine, NYU Langone Health
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: S12-02885
Record Dates: First submitted 2012-10-12; First posted 2012-10-16 (Estimated); Last update posted 2015-09-24 (Estimated); Status verified 2015-09

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

ARMS (2):
- Trans-radial approach (Experimental): Randomized left versus right radial artery approach
  Interventions: Procedure: Randomized left versus right radial artery approach
- Trans-femoral approach (No Intervention): Observational

INTERVENTIONS:
Procedure: Randomized left versus right radial artery approach — Randomized left versus right radial artery approach
  Arms: Trans-radial approach

SUMMARY:
The aim of this study is to measure radiation exposure during coronary angiography (CA) with a trans-radial approach (TRA), specifically comparing access via the left versus right radial artery in patients with suggested clinical predictors of TRA failure/difficult. These predictors include age >70, female gender, height <64 inches, and history of hypertension.The study also aims to determine difficulties encountered during left or right radial access in this specific patient population. A secondary aim is to compare the results of enrolled patients with a registry of patients where femoral access was obtained.

Currently more than 1 million percutaneous coronary interventions (PCI) are performed in the United States annually. There is a growing trend to perform procedures utilizing the TRA due to recent data demonstrating decreased bleeding and access-site complications compared to the femoral approach. However, the TRA approach is also know to be associated with greater radiation exposure compared to the femoral approach. Furthermore, the TRA to catheterization may be difficult in certain populations because of anatomic considerations. Though traditionally completed via canalization of the right radial artery (RRA) due to feasibility with room setup, left radial artery (LRA) access may be superior due to the shorter distance needed to reach the ascending aorta and bypassing the tortuosity of the right subclavian artery. Given the benefits of the TRA, it is important to determine how left versus right radial artery access affects parameters of radiation exposure in addition to procedural difficulty.

This study will be a prospective, randomized study of patients with suggested predictors of TRA failure/difficulty referred for coronary angiography. Patients referred for coronary angiography using the trans-radial approach will be randomly assigned to obtain arterial access via the right or left radial artery. A registry of patients referred for coronary angiography using the trans-femoral approach will be compiled. The primary outcome measure will be radiation exposure as measured by dose area product output from the coronary angiography system. Secondary measures will include the total fluoroscopy time, total dose of radiation, number of catheters used, and incidence of subclavian tortuosity. In addition, procedural complications and success rates will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

Patients referred for cardiac catheterization procedure with 3 out of the following 4 characteristics: age ≥70 years, female gender, hypertensive, and ≤64 inches in height.

Exclusion Criteria:

Patients will be excluded if they 1) underwent prior CABG with utilization of an internal mammary artery, 2) have an abnormal Allen test, 3) require emergency cardiac catheterization, 4) are planned to undergo a staged PCI procedure, 5) do not consent or are unable to give consent, or 6) are participating in another competing study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2012-08; Primary Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Dose area product | During coronary angiography

SECONDARY OUTCOMES:
total fluoroscopy time | during coronary angiography and PCI
total radiation dose | during coronary angiography and PCI
number of catheters used | during coronary angiography
incidence of subclavian tortuosity | during coronary angiography

CONTACTS AND LOCATIONS:
Overall Officials: John Coppola, MD, Principal Investigator — NYU Langone Health; Binita Shah, MD, MS, Principal Investigator — NYU Langone Health
Locations (1):
- New York University Langone Medical Center, New York, New York, United States